CLINICAL TRIAL: NCT03901755
Title: A 24-month Prospective, Non-interventional, International, Multicentre Study to Describe the Real-world Effectiveness and Usage of Alprolix in Patients With Haemophilia B
Brief Title: An International Study to Evaluate the Real-world Effectiveness and Usage of Alprolix in Patients With Haemophilia B
Acronym: B-MORE
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Alprolix-002
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia B
Keywords: Blood Coagulation Disorder; Hematologic Diseases; Coagulation Protein Disorder; Hemorrhagic Disorder; Genetic Diseases, Inborn
MeSH Terms: conditions — Hemophilia B; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — factor IX Fc fusion protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prophylactic patients: Alprolix will be prescribed according to local practice and administered by patients with haemophilia B for prophylactic treatment
  Interventions: Drug: Alprolix
- On demand patients: Alprolix will be prescribed according to local practice and administered by patients with haemophilia B for on-demand treatment
  Interventions: Drug: Alprolix

INTERVENTIONS:
Drug: Alprolix — Extended half-life factor IX product
  Other Names: Eftrenonacog alfa; rFIXFc

SUMMARY:
Alprolix (rFIXFc) is a recombinant extended half-life coagulation factor product. The purpose of this non-interventional study is to describe the real-world usage and effectiveness of Alprolix in the on-demand and prophylactic treatment of haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of haemophilia B
* Have started Alprolix treatment prior to enrolment visit, or at enrolment prescribed treatment with Alprolix irrespective of participation in the study
* Signed and dated informed consent provided by the patient, or the patients legally acceptable representative for patients under the legal age, before any study-related activities are undertaken. Assent should be obtained from paediatric patients according to local regulations.

Exclusion Criteria:

* Participation in an investigational medicinal product trial at enrolment visit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients who present for a routine Clinical visit will be asked to participate in the study by the treating physician at participating haemophilia treatment centres.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Annualised bleeding rate (ABR) | 24 months
  Bleeding episodes assessed according to local practice
Annualised injection frequency | 24 months
  Assessed by prescription
Annualised factor consumption | 24 months
  Assessed by dispensed factor product

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, MD, Study Director — Swedish Orphan Biovitrum
Locations (26):
- Czechia (2):
  - Swedish Orphan Biovitrum Research Site, Brno
  - Swedish Orphan Biovitrum Research Site, Prague
- Greece (2):
  - Swedish Orphan Biovitrum Research Site (Haemophilia Center Aghia Sophia Children's Hospital), Athens
  - Swedish Orphan Biovitrum Research Site (Laikο General Hospital of Athens), Athens
- Swedish Orphan Biovitrum Research Site, Dublin, Ireland
- Italy (6):
  - Swedish Orphan Biovitrum Research Site, Bari
  - Swedish Orphan Biovitrum Research Site, Florence
  - Swedish Orphan Biovitrum Research Site, Genova
  - Swedish Orphan Biovitrum Research Site, Milan
  - Swedish Orphan Biovitrum Research Site, Roma
  - Swedish Orphan Biovitrum Research Site, Turin
- Swedish Orphan Biovitrum Research Site, Oslo, Norway
- Saudi Arabia (2):
  - Swedish Orphan Biovitrum Research Site (King Faisal Hospital adult), Riyadh
  - Swedish Orphan Biovitrum Research Site (King Faisal Hospital pediatric), Riyadh
- Spain (4):
  - Swedish Orphan Biovitrum Research Site (Hospital de Vall d'Hebrón), Barcelona
  - Swedish Orphan Biovitrum Research Site (Hospital Sant Joan de Deu), Barcelona
  - Swedish Orphan Biovitrum Research Site, Murcia
  - Swedish Orphan Biovitrum Research Site, Vigo
- Sweden (4):
  - Swedish Orphan Biovitrum Research Site, Gothenburg
  - Swedish Orphan Biovitrum Research Site, Malmo
  - Swedish Orphan Biovitrum Research Site (Karolinska University Hospital adult), Stockholm
  - Swedish Orphan Biovitrum Research Site (Karolinska University Hospital pediatric), Stockholm
- United Kingdom (4):
  - Swedish Orphan Biovitrum Research Site, Hull
  - Swedish Orphan Biovitrum Research Site, London
  - Swedish Orphan Biovitrum Research Site, Manchester
  - Swedish Orphan Biovitrum Research Site, Oxford

IPD SHARING:
Plan to Share IPD: No